CLINICAL TRIAL: NCT06379178
Title: The Effect of Oral Colostrum Applications Every 2 Hours and 4 Hours In Order to Achieve Trophic Feeding in Preterm Infants
Brief Title: Effect of Oral Colostrum Applications Every 2 Hours and 4 Hours In Order to Achieve Trophic Feeding in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Astri Tantri Indriani, Pediatric neonatology fellow, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6462e56fe8177
Record Dates: First submitted 2024-02-19; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Trophic Feeding; Very Low Birth Weight Baby; Preterm
Keywords: colostrum; very low birth weight; trophic feeding; preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Care 2 Hours (Active Comparator): Oral colostrum application is done every 2 hours
  Interventions: Procedure: Oral colostrum application 2 hours
- Oral care 4 Hours (Active Comparator): Oral colostrum application is done every 4 hours
  Interventions: Procedure: Oral colostrum application 4 hours

INTERVENTIONS:
Procedure: Oral colostrum application 2 hours — Oral colostrum application is an intervention to apply colostrum to oral cavity of subjects. This arm is given oral colostrum application every 2 hours. Colostrum must be from the breastmilk of subject's mother and donor breastmilk is not allowed. Colostrum is treated according to the standard operating procedure of breastmilk storage and preparation of RSUP Dr. Sardjito.
  Arms: Oral Care 2 Hours
Procedure: Oral colostrum application 4 hours — Oral colostrum application is an intervention to apply colostrum to oral cavity of subjects. This arm is given oral colostrum application every 4 hours. Colostrum must be from the breastmilk of subject's mother and donor breastmilk is not allowed. Colostrum is treated according to the standard operating procedure of breastmilk storage and preparation of RSUP Dr. Sardjito.
  Arms: Oral care 4 Hours

SUMMARY:
The goal of this clinical trial is aims to evaluate the effects of applying colostrum orally every 4 and 2 hours in order to achieve trophic feeding in preterm infants. The main question it aims to answer is the optimal frequency of colostrum application that can be applied Participants will be divided by randomization using permutation blocks after meeting the inclusion and exclusion criteria and deemed eligible. These blocks were then randomized using computer software such as Microsoft Excel, determining the sequence for allocation to the control and intervention groups based on the randomization order from the permutation code, every 2 hours and every 4 hours. Researchers will investigate the effects of oropharyngeal colostrum application frequency, every 4 hours and every 2 hours, in order to achieve trophic feeding in preterm infants <34 weeks gestational age.

DETAILED DESCRIPTION:
This study is an experimental research using an open-label Randomized Controlled Trial (RCT) design for a comparative analysis to investigate the effects of oropharyngeal colostrum application frequency, every 4 hours and every 2 hours, in order to achieve trophic feeding in preterm infants <34 weeks gestational age. Inclusion criteria include infants with gestational age <34 weeks, birth weight between 1000-1500 grams, colostrum used was from the mother's own breast milk (not donors' milk), and parents/guardians were willing to participate in the study by signing informed consent. The exclusion criteria involved infants with major congenital abnormalities, infants born to Human Immunodeficiency Virus-positive mothers, infants whose mothers consumed breastfeeding contraindicated drugs, severely ill mothers unable to provide breast milk, and mothers unable to supply breast milk within 48 hours after delivery. The research was conducted after obtaining approval from the Ethics Committee of the Faculty of Medicine, Public Health, and Nursing, UGM, with approval number KE-FK-0811-EC-202.

The sample size was determined using the formula for the independent t-test, requiring a minimum of 14 samples in each group, totaling 28. To account for potential loss to follow-up, the researcher added 10% more samples, resulting in a minimum total of 32 samples. Samples meeting the inclusion and exclusion criteria and deemed eligible underwent randomization using permutation blocks. These blocks were then randomized using computer software such as Microsoft Excel, determining the sequence for allocation to the control and intervention groups based on the randomization order from the permutation code.

The instruments used in this study were the Electronic Medical Record (EMR) from the research subjects and the Case Report Form (CRF). The study necessitated colostrum from the mother's own breast milk, a 1 ml syringe to measure colostrum volume, a tool to facilitate even colostrum application, and a suction catheter to remove excess saliva. The independent variable was the frequency of colostrum application with a categorical variable scale. The dependent variable was the time to achieve trophic feeding with a numerical variable scale, while external variables include necrotizing enterocolitis, sepsis, hsPDA, and gender, represented as categorical variables.

Breast milk expression was initiated within 6 hours post-delivery, adjusted based on the mother's condition. Nurses or doctors assisted with the initial breast milk expression using standard hospital-grade breast pumps or manual methods. Expression was performed by the mother or with the assistance of her spouse every 2-3 hours (eight times per day), with a minimum duration of 10 minutes on each breast. The expressed breast milk was collected in a container, drawn into a 1 ml, 3 ml, or 5 ml syringe depending on the obtained volume, and then labeled for identification. For colostrum application, the nurse took 0.2 ml of colostrum using a 1 ml syringe. Colostrum application prioritized the freshest breast milk, allowing direct administration to the research subject. The remaining breast milk can be used within 2-4 hours at room temperature (16-29 °C) or stored in the refrigerator or freezer according to breast milk storage standards. If frozen, the breast milk should be thawed in the refrigerator before being extracted in the amount of 0.2 ml using a 1 ml syringe for application to the research subject. If stored in the refrigerator, rather than the freezer, 0.2 ml of breast milk should be drawn with a 1 ml syringe, allowed to sit for a designated period (15-30 minutes), and subsequently administered to the research subject.

The administration and preparation of colostrum were performed by a nurse. The nurse conducted an analysis beforehand, following the pre-procedure checklist for colostrum application in the Neonatal Intensive Care Unit (NICU) for each research subject scheduled for colostrum application. If the research subject used mechanical ventilation, the colostrum application procedure was carried out by 2 nurses. Before colostrum application, the oral cavity of the research subject was examined. If excess fluid or saliva was found, suction was performed first, or a sterile gauze was used to remove excess fluid while eliminating dry skin or debris on the lips. Then, with the aid of a 1 ml syringe, colostrum was evenly applied to both right and left cheeks (buccal mucosa), the roof of the mouth, gingival surface, and lips for approximately 1-2 minutes every 2 hours (12 times per day) and every 4 hours (6 times per day). Colostrum in the mouth will be distributed as it mixes with saliva. Colostrum application to the mouth began within 24-48 hours after birth and continued for a total of 5 days.

For research subjects experiencing clinically unstable conditions such as apnea, tachypnea, or desaturation, stabilization was carried out first following the Neonatal Intensive Care Unit (NICU) RSUP Dr. Sardjito Standard Operational Procedure (SOP). After stabilization, colostrum application can be resumed. In cases of feeding intolerance, management was carried out according to the SOP for handling feeding intolerance. If breast milk is available and there are no contraindications to enteral feeding, it can be administered promptly.

Observations of subjects were recorded using the NICU daily monitoring sheet, with detailed notes on various evaluations such as age, days of care, vital signs, feeding intolerance, diagnosis, fluid balance, diuresis, and so forth. Primary research data came from the Case Report Form (CRF) based on the Electronic Medical Record (EMR) and the daily monitoring form in the NICU. The research subjects were prospectively observed, with data being regularly monitored every day until the primary outcomes were achieved, with a maximum observation period of 21 days.

ELIGIBILITY:
Inclusion Criteria:

* infants with gestational age >34 weeks, birth weight 1000-1500 grams, colostrum used was from the mother's own breast milk (not donor's milk), and parents/guardians were willing to participate in the study

Exclusion Criteria:

* infants with major congenital abnormalities ( ), infants born to Human Immunodeficiency Virus-positive mother, infants whose mothers consumed breastfeeding contraindicated drug ( ), severely ill mother unable to provide breast milk, and mothers unable to supply breastmilk within 48 hours after delivery

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2023-02-19 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Days to Achieve Trophic Feeding | Through study completion, an average of 7 days
  Days that subjects achieve and tolerate enteral feeding of10cc per kg of body weight/day

CONTACTS AND LOCATIONS:
Overall Officials: Astri T Indriani, Sp.A, Principal Investigator — Faculty of Medicine, Public Health and Nursing Universitas Gadjah Mada
Locations (1):
- Neonatal Intensive Care Unit RSUP Dr. Sardjito, Sleman, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals should be directed to tantriindrianiastri@gmail.com To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at (Link to be included).